CLINICAL TRIAL: NCT07293273
Title: Impact of Dexmedetomidine and Fentanyl-Propofol Sedation on Peri- and Postprocedural Outcomes in Renal Sympathetic Denervation: A Single-Center Retrospective Study
Brief Title: Procedural Sedation in Renal Sympathetic Denervation
Status: Completed | Type: Observational
Sponsor: Ebru Girgin Dinc (Other)
Responsible Party: Sponsor-Investigator, Ebru Girgin Dinc, M.D., Anesthesiologist, Koşuyolu Kartal Heart Training and Research Hospital
Organization: Koşuyolu Kartal Heart Training and Research Hospital (Other)
Other Study IDs: RSD-S01
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Hypertension, Resistant; Sympathectomy; Conscious Sedation; Procedural Sedation and Analgesia; Dexmedetomidine
Keywords: Dexmedetomidine; Conscious Sedation; Procedural Sedation and Analgesia; sympathectomy; Hypertension, resistant
MeSH Terms: conditions — Hypertension; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal Sympathetic Denervation Patients (Retrospective Cohort): All patients who underwent renal sympathetic denervation for resistant hypertension will be retrospectively included. Within this cohort, patients will be categorized into two subgroups according to sedation regimen:
  Group D: Dexmedetomidine sedation
  Group P: Fentanyl + Propofol sedation
  Comparative analysis will assess peri- and post-procedural safety, hemodynamic stability, and recovery outcomes.

SUMMARY:
This retrospective, single-center study investigates the effects of two different sedation regimens-dexmedetomidine versus fentanyl-propofol-on clinical outcomes in patients undergoing catheter-based renal sympathetic denervation for resistant hypertension. The study focuses on peri-procedural safety, recovery, and overall tolerability of sedation approaches in this interventional setting.

DETAILED DESCRIPTION:
Renal sympathetic denervation has emerged as a therapeutic option for patients with resistant hypertension, yet optimal sedation practices remain unclear. Sedation during catheter-based procedures requires a balance between patient comfort, hemodynamic stability, and minimization of respiratory complications. Dexmedetomidine offers sedative and analgesic effects with minimal respiratory depression, whereas fentanyl-propofol provides rapid, effective sedation but may increase the risk of hemodynamic and respiratory instability. This study retrospectively compares the two strategies by examining intraoperative physiological parameters, complication profiles, and post-procedural recovery measures, aiming to generate evidence that can support anesthesiologists in selecting safer and more effective sedation protocols for this high-risk patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Underwent renal sympathetic denervation for resistant essential hypertension (2023-2024)
* Both male and female

Exclusion Criteria:

* Age <18
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 80 years who underwent renal sympathetic denervation for resistant essential hypertension. Both male and female patients are eligible. Patients younger than 18 years of age and pregnant women are excluded from the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Periprocedural Adverse Events | up to 48 hours
  The primary outcome is a composite of periprocedural adverse events during or immediately after renal sympathetic denervation, defined as the occurrence of any of the following: respiratory depression (SpO₂ <90% ≥1 min or need for airway/ventilation), arrhythmia requiring treatment, need for vasoactive drugs, increase in serum creatinine (KDIGO criteria), or elevation in AST/ALT (>2× baseline or ULN). Patients will be positive if ≥1 event occurs. Comparative analysis will be performed between sedation with dexmedetomidine (Group D) and fentanyl + propofol (Group P).

SECONDARY OUTCOMES:
Dexmedetomidine Dose-Adverse Event Association | up to 48 hours
  Association between total dexmedetomidine dose (µg/kg) and the occurrence of the composite periprocedural adverse event (yes/no).
Propofol Dose-Adverse Event Association | up to 48 hours
  Association between total propofol dose (mg/kg) and the occurrence of the composite periprocedural adverse event (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Ebru GIRGIN DINC, MD, Anesthesiologist, Principal Investigator — Koşuyolu Heart Training and Research Hospital
Locations (1):
- Kosuyolu Heart Training and Research Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol